CLINICAL TRIAL: NCT02678156
Title: Assessment of the Performance of LYoplant® ONlay for Duraplasty. A Non-interventional, Multi-centre Post Market Clinical Follow-up (PMCF) Study.
Brief Title: Assessment of the Performance of LYoplant® ONlay for Duraplasty
Acronym: LYON
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1403
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Craniotomy; Duraplasty; Spinal Surgery
Keywords: Dura mater substitute; Graft; Lyoplant; Lyostypt; Lyoplant onlay; Xenograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LYoplant ONlay: Primary objective of the study is the generation of clinical data in patients receiving Lyoplant® Onlay for dura repair to assess its safety.
  Interventions: Device: Lyoplant Onlay

INTERVENTIONS:
Device: Lyoplant Onlay

SUMMARY:
The aim of this Post Market Clinical Follow-up Study is to collect clinical data on the performance of Lyoplant® Onlay. To assess the performance of the product, various safety and efficacy parameters have been selected.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective cranial or spinal surgery, probably with the need of a duraplasty using Lyoplant® Onlay
* Written informed consent
* Life expectancy > 6 months
* Age > 18 years

Exclusion Criteria:

* Active local or systemic infections
* Open cranial trauma
* Open spina bifida
* Known hypersensitivity to proteins of bovine origin
* Representation by a legal guardian or under involuntary commitment
* Pregnancy
* Participation in another clinical study
* Known primary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Incidence of re-operation because of Cerebrospinal Fluid leakage | until discharge (approximately 1 week)

SECONDARY OUTCOMES:
Incidence of re-operation because of Cerebrospinal Fluid leakage | until follow-up (4 ± 2 months)
Incidence of post operative complications | until discharge (approximately 1 week, 4±2 months)
  Cerebrospinal Fluid leakage, pseudomeningocele, fistulae, infection, meningitis and others
Incidence of cerebral reactions edema, soft tissue swelling, Cerebrospinal Fluid leakage | until discharge (approximately 1 week, 4±2 months)
  detected during routine post operative MRI / CT examinations
Intraoperative handling of the device | Intraoperative
  Intraoperative handling of the device using a questionnaire containing different dimension and a 5 point (1 = excellent, 5 = unacceptable) assessment level (Likert Scale). The following dimensions are assessed:
  * Ease of cutting
  * Needle penetration
  * Adaptation to the tissue
  * Suture retention strength
  * Onlay effect
  * Quality of sealing
  * Thickness
  * Tensile strength
  * Overall satisfaction

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Klinikum Darmstadt, Darmstadt
  - Klinik für Neurochirurgie, Homburg/Saar
  - Klinikum Idar-Oberstein, Idar-Oberstein

IPD SHARING:
Plan to Share IPD: No